CLINICAL TRIAL: NCT00432809
Title: STAMPEDE: Surgical Therapy And Medications Potentially Eradicate Diabetes Efficiently
Brief Title: Advanced Medical Therapy Versus Advanced Medical Therapy Plus Bariatric Surgery for the Resolution of Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Ethicon Endo-Surgery (Industry); LifeScan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EES IIS 19900
Record Dates: First submitted 2007-02-06; First posted 2007-02-08 (Estimated); Results first posted 2013-06-11 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-07

CONDITIONS: Diabetes Mellitus, Type 2; Obesity
Keywords: Diabetes Mellitus, Type 2; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Medical therapy (No Intervention): Intensive medical therapy for diabetes
- Gastric Bypass (Active Comparator): Procedure/Surgery: Bariatric surgery laparoscipic Roux-en-Y Gastric Bypass (RYGB) plus intensive medical therapy
  Interventions: Procedure: Gastric bypass
- Sleeve Gastrectomy (Active Comparator): Procedure/Surgery: Bariatric surgery - laparoscopic sleeve gastrectomy plus intensive medical therapy
  Interventions: Procedure: Sleeve Gastrectomy

INTERVENTIONS:
Procedure: Gastric bypass — Roux-en-Y gastric bypass
  Other Names: RYGB
  Arms: Gastric Bypass
Procedure: Sleeve Gastrectomy — Laparoscopic sleeve gastrectomy
  Other Names: SG
  Arms: Sleeve Gastrectomy

SUMMARY:
The aim of the study is to compare the relative clinical outcomes between advanced medical therapy alone or advanced medical therapy combined with bariatric surgery [either Roux-en-Y gastric bypass (RYGBP) or laparoscopic sleeve gastrectomy] in patients with type 2 diabetes and a body mass index (BMI) between 27 and 43 kg/m2. The study will examine the short and long term effects of each intervention on biochemical resolution of diabetes, diabetic complications, and end-organ damage.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus with HbA1c > 7.0%
* Body mass index > 27 and < 43 kg/m2
* Candidate for general anesthesia

Exclusion Criteria:

* Prior bariatric surgery of any kind
* Cardiovascular conditions including significant coronary artery disease, peripheral vascular disease, uncompensated congestive heart failure, history of stroke, or uncontrolled hypertension
* Kidney disease or chronic renal insufficiency with a creatinine level > 1.8 mg/dl
* Known history of chronic liver disease (except for NAFLD/NASH)
* Gastrointestinal disorders, malabsorptive disorders, or inflammatory bowel disease
* Psychiatric disorders including dementia, active psychosis, severe depression requiring > 2 medications, history of suicide attempts, alcohol or drug abuse within the previous 12 months
* Severe pulmonary disease defined as FEV1 < 50% of predicted value
* Pregnancy

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2007-02; Primary Completion 2016-02 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip R Schauer, MD, Principal Investigator — Director, Bariatric and Metabolic Institute, Cleveland Clinic Foundation
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Background] O'Brien PE, Dixon JB, Laurie C, Skinner S, Proietto J, McNeil J, Strauss B, Marks S, Schachter L, Chapman L, Anderson M. Treatment of mild to moderate obesity with laparoscopic adjustable gastric banding or an intensive medical program: a randomized trial. Ann Intern Med. 2006 May 2;144(9):625-33. doi: 10.7326/0003-4819-144-9-200605020-00005. PMID 16670131
- [Background] Schauer PR, Burguera B, Ikramuddin S, Cottam D, Gourash W, Hamad G, Eid GM, Mattar S, Ramanathan R, Barinas-Mitchel E, Rao RH, Kuller L, Kelley D. Effect of laparoscopic Roux-en Y gastric bypass on type 2 diabetes mellitus. Ann Surg. 2003 Oct;238(4):467-84; discussion 84-5. doi: 10.1097/01.sla.0000089851.41115.1b. PMID 14530719
- [Background] Brethauer SA, Chand B, Schauer PR. Risks and benefits of bariatric surgery: current evidence. Cleve Clin J Med. 2006 Nov;73(11):993-1007. doi: 10.3949/ccjm.73.11.993. PMID 17128540
- [Background] Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):837-53. PMID 9742976
- [Background] Harris MI, Flegal KM, Cowie CC, Eberhardt MS, Goldstein DE, Little RR, Wiedmeyer HM, Byrd-Holt DD. Prevalence of diabetes, impaired fasting glucose, and impaired glucose tolerance in U.S. adults. The Third National Health and Nutrition Examination Survey, 1988-1994. Diabetes Care. 1998 Apr;21(4):518-24. doi: 10.2337/diacare.21.4.518. PMID 9571335
- [Background] Nathan DM. Clinical practice. Initial management of glycemia in type 2 diabetes mellitus. N Engl J Med. 2002 Oct 24;347(17):1342-9. doi: 10.1056/NEJMcp021106. No abstract available. PMID 12397193
- [Background] The relationship of glycemic exposure (HbA1c) to the risk of development and progression of retinopathy in the diabetes control and complications trial. Diabetes. 1995 Aug;44(8):968-83. PMID 7622004
- [Background] Hogan P, Dall T, Nikolov P; American Diabetes Association. Economic costs of diabetes in the US in 2002. Diabetes Care. 2003 Mar;26(3):917-32. doi: 10.2337/diacare.26.3.917. PMID 12610059
- [Derived] Schauer PR, Bhatt DL, Kirwan JP, Wolski K, Aminian A, Brethauer SA, Navaneethan SD, Singh RP, Pothier CE, Nissen SE, Kashyap SR; STAMPEDE Investigators. Bariatric Surgery versus Intensive Medical Therapy for Diabetes - 5-Year Outcomes. N Engl J Med. 2017 Feb 16;376(7):641-651. doi: 10.1056/NEJMoa1600869. PMID 28199805
- [Derived] Schauer PR, Bhatt DL, Kirwan JP, Wolski K, Brethauer SA, Navaneethan SD, Aminian A, Pothier CE, Kim ES, Nissen SE, Kashyap SR; STAMPEDE Investigators. Bariatric surgery versus intensive medical therapy for diabetes--3-year outcomes. N Engl J Med. 2014 May 22;370(21):2002-13. doi: 10.1056/NEJMoa1401329. Epub 2014 Mar 31. PMID 24679060
- [Derived] Kashyap SR, Bhatt DL, Wolski K, Watanabe RM, Abdul-Ghani M, Abood B, Pothier CE, Brethauer S, Nissen S, Gupta M, Kirwan JP, Schauer PR. Metabolic effects of bariatric surgery in patients with moderate obesity and type 2 diabetes: analysis of a randomized control trial comparing surgery with intensive medical treatment. Diabetes Care. 2013 Aug;36(8):2175-82. doi: 10.2337/dc12-1596. Epub 2013 Feb 25. PMID 23439632
- [Derived] Schauer PR, Kashyap SR, Wolski K, Brethauer SA, Kirwan JP, Pothier CE, Thomas S, Abood B, Nissen SE, Bhatt DL. Bariatric surgery versus intensive medical therapy in obese patients with diabetes. N Engl J Med. 2012 Apr 26;366(17):1567-76. doi: 10.1056/NEJMoa1200225. Epub 2012 Mar 26. PMID 22449319

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment began December 2006 and the last patient was enrolled January 2011. Patients were recruited from the Bariatric and Diabetes Outpatient clinic.
Pre-assignment Details: 68 patients screened fail prior to randomization due to not meeting inclusion criteria.
Groups:
- Gastric Bypass: Procedure/Surgery: Bariatric surgery laparoscopic Roux-en-Y Gastric Bypass (RYGB) plus intensive medical therapy
Period: 1 Year Follow-up
Arm/Group | Medical Therapy | Gastric Bypass | Sleeve Gastrectomy
Started | 50 | 50 | 50
Completed | 41 | 50 | 49
Not Completed | 9 | 0 | 1
Not completed — Misses 9 and 12 month visit | 2 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 0 | 1
Period: 2 Year Sub-study
Arm/Group | Medical Therapy | Gastric Bypass | Sleeve Gastrectomy
Started | 20 | 20 | 20
Completed | 17 | 18 | 19
Not Completed | 3 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Medical Therapy | Gastric Bypass | Sleeve Gastrectomy | Total
Number analyzed (Participants) | 50 | 50 | 50 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 50 | 50 | 50 | 150
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.7 (7.4) | 48.3 (8.4) | 47.9 (8.0) | 48.6 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 29 | 39 | 99
  Male | 19 | 21 | 11 | 51
Race/Ethnicity, Customized [Number; unit: participants] — Participants self reported race/ethnicity according to Caucasian, Black/African American, Asian, Hispanic/Latino, American Indian/Alaska Native, Pacific Islander, or Other.
  participants
    Caucasian | 37 | 37 | 36 | 110
    Black/African American | 12 | 13 | 14 | 39
    Asian | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 50 | 150
Duration of diabetes [Mean (Standard Deviation); unit: Years] | 8.9 (5.8) | 8.2 (5.5) | 8.5 (4.8) | 8.5 (5.4)
Use of insulin [Number; unit: participants]
  Insulin dependent | 22 | 22 | 22 | 66
  Non-insulin dependent | 28 | 28 | 28 | 84
body-mass index [Mean (Standard Deviation); unit: kg/m2] | 36.8 (3.0) | 37.0 (3.3) | 36.2 (3.9) | 36.7 (3.4)
Body-mass index < 35 [Number; unit: participants]
  BMI < 35 | 19 | 14 | 18 | 51
  BMI > / = 35 | 31 | 36 | 32 | 99
Body weight [Mean (Standard Deviation); unit: kg] | 106.5 (14.7) | 106.7 (14.8) | 100.8 (16.4) | 104.6 (15.4)
Waist circumference [Mean (Standard Deviation); unit: cm] | 114.5 (9.4) | 116.4 (9.2) | 114.0 (10.4) | 115.0 (9.7)
Fasting glucose [Mean (Standard Deviation); unit: mg/dL] | 169.6 (59.1) | 188.9 (67.6) | 177.6 (70.3) | 178.7 (65.9)
Smoker [Number; unit: Participants]
  Smoker | 15 | 20 | 11 | 46
  Non-smoker | 35 | 30 | 39 | 104
Metabolic syndrome [Number; unit: participants]
  Yes | 46 | 45 | 47 | 138
  No | 4 | 5 | 3 | 12
History of dyslipidemia [Number; unit: participants]
  Yes | 36 | 44 | 40 | 120
  No | 14 | 6 | 10 | 30
History of hypertension [Number; unit: participants]
  Yes | 26 | 35 | 30 | 91
  No | 24 | 15 | 20 | 59
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 137.5 (17.4) | 134.6 (18.7) | 136.2 (18.8) | 136.1 (18.3)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 83.7 (11.5) | 81.8 (10.2) | 82.1 (11.5) | 82.5 (11.0)
High-density lipoprotein cholesterol [Mean (Standard Deviation); unit: mg/dL] | 46.3 (13.2) | 46.2 (13.4) | 44.5 (11.9) | 45.7 (12.8)
Triglycerides [Median (Inter-Quartile Range); unit: mg/dL] | 169.0 [113 to 239] | 167.0 [125 to 257] | 157.0 [119 to 211] | 166.5 [118 to 236]
Diabetic medication - Biguanides [Number; unit: participants]
  Taking Biguanides | 46 | 42 | 42 | 130
  Not taking Biguanides | 4 | 8 | 8 | 20
Diabetes medication - Thiazolidinedione (TZD's) [Number; unit: participants]
  Taking TZD's | 20 | 25 | 17 | 62
  Not taking TZD's | 30 | 25 | 33 | 88
Diabetes medication - Incretin Mimetics [Number; unit: participants]
  Taking Incretin Mimetics | 24 | 19 | 21 | 64
  Not taking Incretin Mimetics | 26 | 31 | 29 | 86
Diabetes medication - Secretagogues [Number; unit: participants]
  Taking Secretagogues | 18 | 17 | 19 | 54
  Not taking Secretagogues | 32 | 33 | 31 | 96
Number of Diabetic Medications [Number; unit: participants]
  0 | 1 | 1 | 1 | 3
  1 | 8 | 10 | 11 | 29
  2 | 11 | 13 | 14 | 38
  3 | 16 | 12 | 13 | 41
  > / = 4 | 14 | 14 | 11 | 39
Cardiovascular medication - Lipid Lowering Agents [Number; unit: participants]
  Taking Lipid Lowering Agent | 41 | 43 | 39 | 123
  Not taking Lipid Lowering Agent | 9 | 7 | 11 | 27
Cardiovascular medication - Beta blocker [Number; unit: participant]
  Taking Beta Blocker | 9 | 9 | 6 | 24
  Not taking Beta Blocker | 41 | 41 | 44 | 126
Cardiovascular medications - ACE Inhibitors or ARB [Number; unit: participant]
  Taking ACE Inhibitor or ARB | 30 | 32 | 25 | 87
  Not taking ACE Inhibitor or ARB | 20 | 18 | 25 | 63
Cardiovascular medication - Anticoagulant [Number; unit: participant]
  Taking Anticoagulants | 26 | 21 | 16 | 63
  Not taking Anticoagulants | 24 | 29 | 34 | 87

OUTCOME MEASURES:

1. Primary Outcome: Success Rate of Biochemical Resolution of Diabetes at 12 Months as Measured by HbA1c ≤ 6%.
Description: The proportion of subjects with a glycated hemoglobin level of 6% or less(with or without diabetes medications) 12 months after randomization (baseline measure).
Time Frame: 1 year
Population: Modified intent-to-treat (ITT) population consists of all randomized patients that initiate treatment (surgery for those randomized to surgery and medical treatment for those randomized to medical treatment). All analyses conducted in the modified ITT population. Primary analysis also conducted in per protocol population as a sensitivity analysis.
Measure: Number; unit: participants
Arm/Group | Medical Therapy | Gastric Bypass | Sleeve Gastrectomy
Number analyzed (Participants) | 41 | 50 | 49
participants | 5 | 21 | 18
Statistical Analysis 1: Comparison: Medical Therapy vs Gastric Bypass; Test type: Superiority or Other; p = 0.002, Chi-squared
Statistical Analysis 2: Comparison: Medical Therapy vs Sleeve Gastrectomy; Test type: Superiority or Other; p = 0.008, Chi-squared
Statistical Analysis 3: Comparison: Gastric Bypass vs Sleeve Gastrectomy; Test type: Superiority or Other; p = 0.59, Chi-squared — Not adjusted for multiple comparisons

2. Secondary Outcome: Changes in Specific Metabolic Parameters (Insulin Secretion and Resistance).
Time Frame: 1, 2, and 5 years
Reporting Status: Not Posted

3. Secondary Outcome: Changes in Obesity-related Comorbidities (Blood Pressure, Dyslipidemia), Quality of Life, and Hospitalizations.
Time Frame: 1, 2, and 5 years
Reporting Status: Not Posted

4. Secondary Outcome: The Cost-effectiveness of Each Program and the Side Effects and /or Complications.
Time Frame: 1, 2, and 5 years.
Reporting Status: Not Posted

5. Secondary Outcome: Change in Glycated Hemoglobin (HbA1c)
Description: Change in glycated hemoglobin(HbA1c)from baseline in percentage points / percent change
Time Frame: 1 year - baseline
Population: Modified intent-to-treat population consists of all randomized patients that initiate treatment (surgery for those randomized to surgery and medical treatment for those randomized to medical treatment). All analyses conducted in the modified ITT population. Primary analysis also conducted in per protocol population as a sensitivity analysis.
Measure: Mean (Standard Deviation); unit: percentage points of glycated hemoglobin
Arm/Group | Medical Therapy | Gastric Bypass | Sleeve Gastrectomy
Number analyzed (Participants) | 41 | 50 | 49
percentage points of glycated hemoglobin | -1.4 (1.5) | -2.9 (1.6) | -2.9 (1.8)
Statistical Analysis 1: Comparison: Medical Therapy vs Gastric Bypass; Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Medical Therapy vs Sleeve Gastrectomy; Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 3: Comparison: Gastric Bypass vs Sleeve Gastrectomy; Test type: Superiority or Other; p = 0.85, ANOVA

6. Secondary Outcome: Fasting Plasma Glucose
Description: Fasting Plasma Glucose measured in mg/dL.
Time Frame: 1 year
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Medical Therapy | Gastric Bypass | Sleeve Gastrectomy
Number analyzed (Participants) | 41 | 50 | 49
mg/dL | 120 [97 to 154] | 99 [83 to 121] | 97 [84 to 114]
Statistical Analysis 1: Comparison: Medical Therapy vs Gastric Bypass; Test type: Superiority or Other; p = 0.004, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Medical Therapy vs Sleeve Gastrectomy; Test type: Superiority or Other; p = 0.003, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Gastric Bypass vs Sleeve Gastrectomy; Test type: Superiority or Other; p = 0.86, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Glycated Hemoglobin (HbA1c)
Description: Mean glycated hemoglobin (HbA1c) at 12 months for each of the 3 groups, in percentage points
Time Frame: 1 year
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage points of glycated hemoglobin
Arm/Group | Medical Therapy | Gastric Bypass | Sleeve Gastrectomy
Number analyzed (Participants) | 41 | 50 | 49
percentage points of glycated hemoglobin | 7.5 (1.8) | 6.4 (0.9) | 6.6 (1.0)
Statistical Analysis 1: Comparison: Medical Therapy vs Gastric Bypass; Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Medical Therapy vs Sleeve Gastrectomy; Test type: Superiority or Other; p = 0.003, ANOVA
Statistical Analysis 3: Comparison: Gastric Bypass vs Sleeve Gastrectomy; Test type: Superiority or Other; p = 0.23, ANOVA

8. Primary Outcome: Success Rate of Biochemical Resolution of Diabetes at 12 Months as Measured by HbA1c ≤ 6% With no Diabetes Medications
Description: The proportion of subjects with a glycated hemoglobin level of 6% or less(without diabetes medications) 12 months after randomization.
Time Frame: 1 year
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Medical Therapy | Gastric Bypass | Sleeve Gastrectomy
Number analyzed (Participants) | 41 | 50 | 49
participants | 0 | 21 | 13
Statistical Analysis 1: Comparison: Medical Therapy vs Gastric Bypass; Medical Therapy vs. Gastric Bypass; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: Medical Therapy vs Sleeve Gastrectomy; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 3: Comparison: Gastric Bypass vs Sleeve Gastrectomy; Test type: Superiority or Other; p = 0.10, Chi-squared

9. Secondary Outcome: Body Weight
Description: Body weight in kilograms (kg) measured at 12 months
Time Frame: 1 year
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Medical Therapy | Gastric Bypass | Sleeve Gastrectomy
Number analyzed (Participants) | 41 | 50 | 49
kg | 99.0 (16.4) | 77.3 (13.0) | 75.5 (12.9)
Statistical Analysis 1: Comparison: Medical Therapy vs Gastric Bypass; Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Medical Therapy vs Sleeve Gastrectomy; Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 3: Comparison: Gastric Bypass vs Sleeve Gastrectomy; Test type: Superiority or Other; p = 0.02, ANOVA

10. Secondary Outcome: Change in Body Weight From Baseline
Description: Mean change in body weight from baseline measured in kilograms (kg)
Time Frame: 1 year
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Medical Therapy | Gastric Bypass | Sleeve Gastrectomy
Number analyzed (Participants) | 41 | 50 | 49
kg | -5.4 (8.0) | -29.4 (8.9) | -25.1 (8.5)
Statistical Analysis 1: Comparison: Medical Therapy vs Gastric Bypass; Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Medical Therapy vs Sleeve Gastrectomy; Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 3: Comparison: Gastric Bypass vs Sleeve Gastrectomy; Test type: Superiority or Other; p = 0.02, ANOVA

11. Secondary Outcome: Body Mass Index (BMI)
Description: Body Mass Index (BMI) at 12 months measured as kg/m2
Time Frame: 1 year
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Medical Therapy | Gastric Bypass | Sleeve Gastrectomy
Number analyzed (Participants) | 41 | 50 | 49
kg/m2 | 34.4 (3.7) | 26.8 (3.2) | 27.2 (3.5)
Statistical Analysis 1: Comparison: Medical Therapy vs Gastric Bypass; Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Medical Therapy vs Sleeve Gastrectomy; Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 3: Comparison: Gastric Bypass vs Sleeve Gastrectomy; Test type: Superiority or Other; p = 0.61, ANOVA

12. Secondary Outcome: Change in Body Mass Index (BMI)
Description: Change in Body Mass Index (BMI) at 12 months, measured in kg/m2
Time Frame: 1 year
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Medical Therapy | Gastric Bypass | Sleeve Gastrectomy
Number analyzed (Participants) | 41 | 50 | 49
kg/m2 | -1.9 (2.9) | -10.2 (3.1) | -9.0 (2.7)
Statistical Analysis 1: Comparison: Medical Therapy vs Gastric Bypass; Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Medical Therapy vs Sleeve Gastrectomy; Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 3: Comparison: Gastric Bypass vs Sleeve Gastrectomy; Test type: Superiority or Other; p = 0.03, ANOVA

13. Secondary Outcome: Change in Systolic Blood Pressure (SBP)
Description: Change in Systolic Blood Pressure (SBP) at 12 months
Time Frame: 1 year
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Medical Therapy | Gastric Bypass | Sleeve Gastrectomy
Number analyzed (Participants) | 41 | 50 | 49
mm Hg | -3.9 (14.7) | -2.4 (18.7) | -5.1 (17.0)
Statistical Analysis 1: Comparison: Medical Therapy vs Gastric Bypass; Test type: Superiority or Other; p = 0.87, ANOVA
Statistical Analysis 2: Comparison: Medical Therapy vs Sleeve Gastrectomy; Test type: Superiority or Other; p = 0.67, ANOVA
Statistical Analysis 3: Comparison: Gastric Bypass vs Sleeve Gastrectomy; Test type: Superiority or Other; p = 0.46, ANOVA

14. Secondary Outcome: Change in High-density Lipoprotein (HDL)
Description: Percent change in high-density lipoprotein (HDL) at 12 months
Time Frame: 1 year
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Medical Therapy | Gastric Bypass | Sleeve Gastrectomy
Number analyzed (Participants) | 41 | 50 | 49
mg/dL | 11.3 (25.7) | 28.5 (22.7) | 28.4 (21.9)
Statistical Analysis 1: Comparison: Medical Therapy vs Gastric Bypass; Test type: Superiority or Other; p = 0.001, ANOVA
Statistical Analysis 2: Comparison: Medical Therapy vs Sleeve Gastrectomy; Test type: Superiority or Other; p = 0.001, ANOVA
Statistical Analysis 3: Comparison: Gastric Bypass vs Sleeve Gastrectomy; Test type: Superiority or Other; p = 0.98, ANOVA

15. Secondary Outcome: Change in Triglycerides
Description: Median percent change in triglycerides at 12 months from baseline measure
Time Frame: 1 year
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Medical Therapy | Gastric Bypass | Sleeve Gastrectomy
Number analyzed (Participants) | 41 | 50 | 49
mg/dL | -14 [-40 to 3] | -44 [-65 to -16] | -42 [-56 to 0]
Statistical Analysis 1: Comparison: Medical Therapy vs Gastric Bypass; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Medical Therapy vs Sleeve Gastrectomy; Test type: Superiority or Other; p = 0.08, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Gastric Bypass vs Sleeve Gastrectomy; Test type: Superiority or Other; p = 0.17, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Change in High-sensitivity C-reactive Protein (Hs-CRP)
Description: Median percent change in high-sensitivity C-reactive protein (hs-CRP)from baseline at 12 months
Time Frame: 1 year
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Medical Therapy | Gastric Bypass | Sleeve Gastrectomy
Number analyzed (Participants) | 41 | 50 | 49
mg/L | -33.2 [-71 to 0] | -84 [-91 to -59] | -80 [-90 to -63]
Statistical Analysis 1: Comparison: Medical Therapy vs Gastric Bypass; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Medical Therapy vs Sleeve Gastrectomy; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Gastric Bypass vs Sleeve Gastrectomy; Test type: Superiority or Other; p = 0.59, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: Diabetes Medication - Use of Insulin
Description: Number of participants taking insulin at 12 months
Time Frame: 1 year
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Medical Therapy | Gastric Bypass | Sleeve Gastrectomy
Number analyzed (Participants) | 41 | 50 | 49
participants | 15 | 2 | 4
Statistical Analysis 1: Comparison: Medical Therapy vs Gastric Bypass; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: Medical Therapy vs Sleeve Gastrectomy; Test type: Superiority or Other; p = 1.001, Chi-squared
Statistical Analysis 3: Comparison: Gastric Bypass vs Sleeve Gastrectomy; Test type: Superiority or Other; p = 0.68, Chi-squared

18. Secondary Outcome: Diabetes Medication - Use of Biguanides
Description: Number of participants taking Biguanides at 12 months
Time Frame: 1 year
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Medical Therapy | Gastric Bypass | Sleeve Gastrectomy
Number analyzed (Participants) | 41 | 50 | 49
participants | 38 | 10 | 19
Statistical Analysis 1: Comparison: Medical Therapy vs Gastric Bypass; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: Medical Therapy vs Sleeve Gastrectomy; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 3: Comparison: Gastric Bypass vs Sleeve Gastrectomy; Test type: Superiority or Other; p = 0.05, Chi-squared

19. Secondary Outcome: Diabetes Medication - Use of Thiazolidinedione
Description: Number of participants using thiazolidinedione at 12 months
Time Frame: 1 year
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Medical Therapy | Gastric Bypass | Sleeve Gastrectomy
Number analyzed (Participants) | 41 | 50 | 49
participants | 20 | 0 | 5
Statistical Analysis 1: Comparison: Medical Therapy vs Gastric Bypass; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: Medical Therapy vs Sleeve Gastrectomy; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 3: Comparison: Gastric Bypass vs Sleeve Gastrectomy; Test type: Superiority or Other; p = 0.06, Chi-squared

20. Secondary Outcome: Diabetes Medication - Use of Incretin Mimetics
Description: Number of participants taking Incretin Mimetics
Time Frame: 1 year
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Medical Therapy | Gastric Bypass | Sleeve Gastrectomy
Number analyzed (Participants) | 41 | 50 | 49
participants | 34 | 1 | 10
Statistical Analysis 1: Comparison: Medical Therapy vs Gastric Bypass; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: Medical Therapy vs Sleeve Gastrectomy; Test type: Superiority or Other; p = 0.005, Chi-squared
Statistical Analysis 3: Comparison: Gastric Bypass vs Sleeve Gastrectomy; Test type: Superiority or Other; p = 0.004, Chi-squared

21. Secondary Outcome: Diabetes Medication - Use of Secretagogue
Description: Number of participants taking Secretagogues at 12 months
Time Frame: 1 year
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Medical Therapy | Gastric Bypass | Sleeve Gastrectomy
Number analyzed (Participants) | 41 | 50 | 49
participants | 10 | 1 | 5
Statistical Analysis 1: Comparison: Medical Therapy vs Gastric Bypass; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: Medical Therapy vs Sleeve Gastrectomy; Test type: Superiority or Other; p = 0.06, Chi-squared
Statistical Analysis 3: Comparison: Gastric Bypass vs Sleeve Gastrectomy; Test type: Superiority or Other; p = 0.20, Chi-squared

22. Secondary Outcome: Cardiovascular Medications - Lipid Lowering Agents
Description: Number of participants taking Lipid lowering agents at 12 months
Time Frame: 1 year
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Medical Therapy | Gastric Bypass | Sleeve Gastrectomy
Number analyzed (Participants) | 41 | 50 | 49
participants | 36 | 13 | 19
Statistical Analysis 1: Comparison: Medical Therapy vs Gastric Bypass; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: Medical Therapy vs Sleeve Gastrectomy; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 3: Comparison: Gastric Bypass vs Sleeve Gastrectomy; Test type: Superiority or Other; p = 0.20, Chi-squared

23. Secondary Outcome: Cardiovascular Medications - Beta Blocker
Description: Number of participants taking Beta Blockers at 12 months
Time Frame: 1 year
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Medical Therapy | Gastric Bypass | Sleeve Gastrectomy
Number analyzed (Participants) | 41 | 50 | 49
participants | 5 | 9 | 3
Statistical Analysis 1: Comparison: Medical Therapy vs Gastric Bypass; Test type: Superiority or Other; p = 0.48, Chi-squared
Statistical Analysis 2: Comparison: Medical Therapy vs Sleeve Gastrectomy; Test type: Superiority or Other; p = 0.46, Chi-squared
Statistical Analysis 3: Comparison: Gastric Bypass vs Sleeve Gastrectomy; Test type: Superiority or Other; p = 0.06, Chi-squared

24. Secondary Outcome: Cardiovascular Medications - Angiotensin-converting Enzyme (ACE Inhibitor) or Angiotensin-receptor Blocker (ARB)
Description: Number of participants taking Angiotensin-converting enzyme (ACE Inhibitor) or Angiotensin-receptor blocker (ARB) at 12 months
Time Frame: 1 year
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Medical Therapy | Gastric Bypass | Sleeve Gastrectomy
Number analyzed (Participants) | 41 | 50 | 49
participants | 26 | 9 | 11
Statistical Analysis 1: Comparison: Medical Therapy vs Gastric Bypass; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: Medical Therapy vs Sleeve Gastrectomy; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 3: Comparison: Gastric Bypass vs Sleeve Gastrectomy; Test type: Superiority or Other; p = 0.62, Chi-squared

25. Secondary Outcome: Cardiovascular Medications - Anticoagulants
Description: Number of participants taking anticoagulants at 12 months
Time Frame: 1 year
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Medical Therapy | Gastric Bypass | Sleeve Gastrectomy
Number analyzed (Participants) | 41 | 50 | 49
participants | 24 | 1 | 8
Statistical Analysis 1: Comparison: Medical Therapy vs Gastric Bypass; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: Medical Therapy vs Sleeve Gastrectomy; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 3: Comparison: Gastric Bypass vs Sleeve Gastrectomy; Test type: Superiority or Other; p = 0.03, Chi-squared

ADVERSE EVENTS:
Time Frame: 1 year
Description: Subjects systematically assessed every 3 months during routine study visits, or sooner if an event occurred.
  Number of Medical Therapy subjects (43) includes 2 subjects that had an event and withdrew consent prior to their 9 month visit. 7 subjects withdrew immediately after randomization.
  1 Sleeve Gastrectomy subject withdrew prior to surgery.
Arm/Group | Medical Therapy | Gastric Bypass | Sleeve Gastrectomy
Serious Adverse Events (participants affected / at risk) | 4/43 | 16/50 | 7/49
Other Adverse Events (participants affected / at risk) | 42/43 | 48/50 | 49/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medical Therapy (N=43) | Gastric Bypass (N=50) | Sleeve Gastrectomy (N=49)
Intravenous treatment for dehydration (Surgical and medical procedures) | 0 (0) | 4 (4) | 2 (2) — Intravenous treatment for dehydration requiring hospitalization
Reoperation (Surgical and medical procedures) | 0 (0) | 3 (3) | 1 (1)
Transfusion (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1)
Hemoglobin decrease > / = 5 g/dl (Investigations) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal leak (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Transient renal insufficiency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (2) | 0 (0)
Arrhythmia or palpitations (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Ketoacidosis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Kidney stone (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hernia (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medical Therapy (N=43) | Gastric Bypass (N=50) | Sleeve Gastrectomy (N=49)
IV Treatment for Dehydration (Surgical and medical procedures) | 1 (1) | 6 (8) | 4 (4)
Reflux Disease - GERD (Surgical and medical procedures) | 1 (1) | 4 (4) | 7 (7)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 8 (12) | 8 (9)
Constipation (Gastrointestinal disorders) | 6 (7) | 9 (9) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 4 (4) | 3 (3)
Nausea (Gastrointestinal disorders) | 4 (4) | 7 (12) | 8 (8)
Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (9) | 8 (8)
Fatty Liver (Hepatobiliary disorders) | 0 (0) | 26 (27) | 24 (25)
Infection Not Requiring Antibiotics (Infections and infestations) | 3 (3) | 3 (3) | 2 (2)
Infections Requiring Antibiotics (Infections and infestations) | 7 (9) | 6 (10) | 5 (6)
Viral Flu (Infections and infestations) | 12 (14) | 5 (6) | 9 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 6 (6) | 3 (4)
Fatigue (Musculoskeletal and connective tissue disorders) | 3 (4) | 4 (4) | 3 (3)
Foot pain (Musculoskeletal and connective tissue disorders) | 5 (7) | 3 (3) | 3 (3)
Hand pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2) | 1 (1)
Hip pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (7) | 2 (2)
Knee pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 4 (4)
Muscle pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2) | 4 (4)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 5 (5) | 6 (6)
Headache (Nervous system disorders) | 2 (3) | 2 (2) | 4 (5)
Numbness (Nervous system disorders) | 3 (3) | 3 (3) | 2 (2)
Vertigo / Dizziness (Nervous system disorders) | 3 (3) | 10 (10) | 9 (9)
Depression (Psychiatric disorders) | 7 (7) | 2 (2) | 6 (6)
UTI (Urinary Tract Infection) (Renal and urinary disorders) | 5 (5) | 2 (2) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 3 (3)
Upper Respiratory Infection - Bacterial (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (6) | 5 (7)
Upper Respiratory Infection - Viral (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 6 (8) | 5 (5)
Alopecia / hair loss (Skin and subcutaneous tissue disorders) | 3 (3) | 20 (21) | 18 (18)

LIMITATIONS AND CAVEATS:
Important limitations in the primary endpoint and 1 year outcomes are the short duration of follow-up (12 months), the study occurred at a single-center and the open-label nature of the study (subjects were not blinded to treatment).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes